CLINICAL TRIAL: NCT04256512
Title: Cryotherapy to Prevent Taxane-Induced Sensory Neuropathy of the Hands and Feet
Brief Title: Cryotherapy for the Prevention of Taxane-Induced Sensory Neuropathy of the Hands and Feet in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-008929; NCI-2021-02755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-008929 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prevention (Elasto Gel Therapy Mittens and Foot Wraps) (Experimental): Patients wear Elasto Gel Therapy Mittens and Foot Wraps on both hands and feet 15 minutes prior to each infusion, during the entire infusion, and for 15 minutes after the completion of each infusion during their three months of treatment.
  Interventions: Device: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Device: Medical Device Usage and Evaluation — Wear Elasto Gel Therapy Mittens and Foot Wraps
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial investigates the effect and tolerability of cryotherapy and to evaluate whether they can prevent or improve taxane-induced sensory peripheral neuropathy in breast cancer patients. Cryosurgery, also known as cryoablation or cryotherapy, kills tumor cells by freezing them. Patients receiving cryotherapy during infusion of taxane therapy may have lower incidence of peripheral neuropathy, better physical function, and higher quality of life as compared to patients previously reported in literature.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the efficacy and tolerability of cryotherapy (Elasto Gel frozen mittens and foot wraps) and to evaluate whether they can prevent or ameliorate taxane-induced sensory peripheral neuropathy.

OUTLINE:

Patients wear Elasto Gel Therapy Mittens and Foot Wraps on both hands and feet 15 minutes prior to each infusion, during the entire infusion, and for 15 minutes after the completion of each infusion during their three months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age with a diagnosis of breast cancer
* Patients receiving 12-18 weeks of chemotherapy with a taxane-based regimen (4 cycles of weekly x 3 paclitaxel or 4-6 cycles of docetaxel every 3 weeks)
* Absence of sensory peripheral neuropathy, skin or nail disorders at the start of treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Ability to complete questionnaires by themselves or with assistance
* Ability to give signed informed consent

Exclusion Criteria:

* History of prior sensory/motor peripheral neuropathy from any cause
* History of prior Raynaud's phenomenon
* History of cryoglobulinemia
* Active peripheral vascular disease
* Cold intolerance
* Prior exposure to neurotoxic chemotherapy in the last 10 years
* Hand-foot syndrome
* Tumor metastasis in bone, soft tissue, or skin of the hands or feet
* Absence of one or more fingers or toes
* Prior exposure to taxane chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Advani, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single arm non-randomized study was conducted at Mayo Clinic in Florida. Participants included early breast cancer patients who underwent standard of care chemotherapy and who had Eastern Cooperative Oncology Group (ECOG) performance status 0-2 with no sensory peripheral neuropathy at study entry. Patients with metastatic breast cancer, Raynaud's and peripheral vascular disease, cryoglobulinemia, cold intolerance, prior exposure to neurotoxic or taxane chemotherapy were excluded.
Period: Overall Study
Arm/Group | Prevention (Elasto Gel Therapy Mittens and Foot Wraps)
Started | 94
Completed | 93
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Elasto Gel Therapy Mittens and Foot Wraps)
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 14
Age, Continuous [Median (Standard Deviation); unit: years] | 54 (12.270)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Pacific Islander | 0
  Black or African American | 22
  White | 62
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Chemotherapy Induced Peripheral Neuropathy (CIPN)
Description: Number of subjects to experience chemotherapy induced peripheral neuropathy (CIPN).
Time Frame: During chemotherapy (baseline), after chemotherapy (1 week post baseline), at 3 month follow up
Population: Adults ages 18 and older with diagnosis of breast cancer undergoing 3 months of taxane based chemotherapy [4 cycles of weekly paclitaxel (1 cycle = 3 weeks) or docetaxel every 3 weeks x 4-6 cycles].
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Elasto Gel Therapy Mittens and Foot Wraps)
Number analyzed (Participants) | 93
Participants
  During chemotherapy | 41
  After chemotherapy: number analyzed (Participants) | 82
  After chemotherapy | 30
  3 month follow up: number analyzed (Participants) | 80
  3 month follow up | 25

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected prior to each cycle of chemo, at the end of each cycle, and 3 months after chemotherapy.
Description: Patients were evaluated for chemotherapy induced peripheral neuropathy (CIPN).
Arm/Group | Prevention (Elasto Gel Therapy Mittens and Foot Wraps)
All-Cause Mortality (participants affected / at risk) | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 41/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prevention (Elasto Gel Therapy Mittens and Foot Wraps) (N=93)
Neuropathy during chemotherapy (Grade 1) (Nervous system disorders) | 41 (41)
Neuropathy after chemotherapy (Grade 1) (Nervous system disorders) | 28/82 (28) — 11 patients withdrew prior to the 'neuropathy after chemo' visit
Neuropathy after chemotherapy (Grade 2) (Nervous system disorders) | 2/82 (2) — 11 patients withdrew prior to the 'neuropathy after chemo' visit
Neuropathy at 3 month follow up (Grade 1) (Nervous system disorders) | 19/80 (19) — 13 patients withdrew prior to the 'neuropathy at 3-month follow-up' visit
Neuropathy at 3 month follow up (Grade 2) (Nervous system disorders) | 6/80 (6) — 13 patients withdrew prior to the 'neuropathy at 3-month follow-up' visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT04256512/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04256512/ICF_001.pdf